CLINICAL TRIAL: NCT00000862
Title: A Phase I Trial of the Pharmacokinetics and Tolerance of Oral Zidovudine Administered to HIV-1 Infected Pregnant Women During Labor and Delivery
Brief Title: A Study of Zidovudine During Labor and Delivery in HIV-Infected Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 324; 11298 (Registry Identifier: DAIDS ES Registry Number); PACTG 324
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Administration, Oral; Zidovudine; Delivery; Labor; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To obtain a pharmacokinetic profile of oral ZDV and to determine whether the oral administration of Zidovudine (ZDV) during labor and delivery will provide a similar profile to that obtained with the use of IV ZDV in ACTG 082. To evaluate the tolerance of oral ZDV in this population, defined as the ability to take oral doses and lack of vomiting within 30 minutes of receiving oral study doses.

The worldwide use of constant intrapartum ZDV infusions to prevent transmission is not practical or feasible. Approximately 18% of the women in the ACTG 076 trial missed their IV ZDV infusions, even at experienced ACTG sites. There is an urgent need to establish a more practical method of delivering ZDV during labor and delivery that, at minimum, will approximate the rate of ZDV administration utilized in ACTG 082. In the future, this would enable women to start an intensive ZDV regimen during early labor, even prior to reaching the hospital.

DETAILED DESCRIPTION:
The worldwide use of constant intrapartum ZDV infusions to prevent transmission is not practical or feasible. Approximately 18% of the women in the ACTG 076 trial missed their IV ZDV infusions, even at experienced ACTG sites. There is an urgent need to establish a more practical method of delivering ZDV during labor and delivery that, at minimum, will approximate the rate of ZDV administration utilized in ACTG 082. In the future, this would enable women to start an intensive ZDV regimen during early labor, even prior to reaching the hospital.

Cohort 1: Women in active labor receive 3 doses of oral ZDV 3 hours apart followed by PK sampling. After PK sampling post 3rd oral dose, or at 8 cm dilation (whichever comes first), women receive IV ZDV until delivery. The cord blood will be analyzed for serum ZDV PK levels and the infant's infection status will be determined. If the dose of ZDV is adequate to achieve targeted maternal serum drug levels in Cohort 1 and if oral dosing is tolerated in this cohort, Cohort 2 will begin enrollment. [AS PER AMENDMENT 08/03/01: Cohort 1 has been completed and only Cohort 2 is open for enrollment.] Cohort 2: [AS PER AMENDMENT 08/03/01: Women in active labor receive initial loading dose of oral ZDV, then another dose of oral ZDV 3 hours later, both doses followed by PK sampling. After PK sampling post second oral dose, or at 8 cm dilation (whichever comes first), woman receives IV ZDV until delivery. The cord blood will not be analyzed for serum ZDV PK levels and the infant's infection status will be determined.]

ELIGIBILITY:
Inclusion Criteria

A woman may be eligible for this study if:

* She is HIV-positive.
* She is at least 34 weeks pregnant.
* She has a history of at least 4 weeks of continuous oral ZDV during her current pregnancy and tolerated it well.
* She has given consent for her newborn to participate in this study. (The father must also give consent if he is available after reasonable attempts to contact him. A woman under 18 needs the consent of a parent or legal guardian for her and her infant to participate.)

Exclusion Criteria

A woman will not be eligible for this study if:

* She is taking part in another study of HIV treatment during pregnancy.
* Her infant has a life-threatening illness indicated in an ultrasound.
* Her infant does not appear to be growing normally in the womb.
* She has a cesarean section.
* She has abnormal blood test results.
* She has severe nausea, vomiting, or other problems of the stomach and intestines at the time of study entry.
* She has an active opportunistic (AIDS-related) infection or other serious infection at the time of study entry.
* The study staff cannot find a usable vein.
* The study doctor feels that she cannot take drugs by mouth.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, Study Chair; Pamela Boyer, Study Chair
Locations (11):
- United States (10):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Univ of California, San Francisco, San Francisco, California
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
- San Juan City Hosp, San Juan, Puerto Rico